CLINICAL TRIAL: NCT02140944
Title: IMPAACT P1107: Cord Blood Transplantation With CCR5Δ32 Donor Cells in HIV-1 Infected Subjects Who Require Bone Marrow Transplantation for Any Indication and Its Observed Effects on HIV-1 Persistence
Brief Title: IMPAACT P1107: Effects of Cord Blood Transplantation With CCR5Δ32 Donor Cells on HIV Persistence
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1107; UM1AI068632 (NIH); UM1AI068616 (NIH); UM1AI106716 (NIH)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: HIV Infection
Keywords: Cord blood transplantation; CCR5Δ32; HIV cure
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For consenting participants, blood and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-Transplant Cohort: HIV-1 infected participants, enrolled prior to transplant, who receive a heterozygous or homozygous CCR∆32 cord blood transplant
- Post-Transplant Cohort: HIV-1 infected participants, enrolled within 2 years after transplant, who receive a homozygous CCR∆32 cord blood transplant

SUMMARY:
IMPAACT P1107 will describe the outcomes of HIV-infected persons, ages 12 months and older, who undergo transplantation with CCR5Δ32 cord blood stem cells for treatment of cancer, hematopoietic disease, or other underlying disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection
* 12 months of age or older
* Willing to provide written informed consent
* Pre-Transplant Cohort: Underlying disease appropriate for stem cell transplant, as determined by the transplant team as part of standard of care.
* Pre-Transplant Cohort: Availability of an appropriately matched (as determined by the transplant center) CCR5Δ32 cord blood unit (homozygous or heterozygous) and intention to proceed with transplantation. NOTE: Double cord transplants are allowed. If a double cord is used, at least one cord blood unit should be CCR5∆32 (homozygous or heterozygous).
* Pre-Transplant Cohort: Received a CCR5Δ32 homozygous cord blood or bone marrow transplant within the last two years.

Exclusion Criteria:

• Received, or planning to receive, more than one CCR5Δ32 homozygous cord blood or bone marrow transplant.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-1 infected children and adults who undergo cord blood stem cell transplantation for treatment of cancer, hematopoietic disease, or other underlying disease
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Survival | Through 5 years post-transplant
  Survival and event-free survival at 100 days, Week 26, Week 52, and then every six months until five years post-transplant
Graft versus host disease | Through 5 years post-transplant
  Graft versus host disease
Engraftment | Through 5 years post-transplant
  Chimerism (≥ 98% of blood cells bearing CCR5∆32) and time to hematopoietic cell and immune recovery
HIV DNA level | Through 5 years post-transplant
  HIV-1 proviral DNA levels in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bryson, MD, Study Chair — University of California, Los Angeles
Locations (1):
- Weill Cornell Uptown Clinical Research Site (7803), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Hsu J, Van Besien K, Glesby MJ, Pahwa S, Coletti A, Warshaw MG, Petz L, Moore TB, Chen YH, Pallikkuth S, Dhummakupt A, Cortado R, Golner A, Bone F, Baldo M, Riches M, Mellors JW, Tobin NH, Browning R, Persaud D, Bryson Y; International Maternal Pediatric Adolescent AIDS Clinical Trials Network (IMPAACT) P1107 Team. HIV-1 remission and possible cure in a woman after haplo-cord blood transplant. Cell. 2023 Mar 16;186(6):1115-1126.e8. doi: 10.1016/j.cell.2023.02.030. PMID 36931242
- See also: Study website — http://www.impaactnetwork.org/studies/P1107.asp